CLINICAL TRIAL: NCT02602353
Title: A Phase 2, Randomized, Double-Blind, Parallel-Group and Placebo-Controlled Pilot Study to Assess the Safety and Efficacy of a New Pain Patch Versus Placebo and No Treatment for the Treatment of Delayed Onset Muscle Soreness (DOMS)
Brief Title: Pilot Study Comparing the Efficacy and Safety of a New Pain Patch and Placebo in Delayed Onset Muscle Soreness (DOMS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lead Chemical Co., Ltd. (Industry)
Collaborators: Cardinal Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEAD-PhII-050
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Delayed Onset Muscle Soreness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Loxoprofen Pain Patch (Experimental): One Active Pain Patch containing loxoprofen applied once daily for 3 days
  Interventions: Drug: Loxoprofen Pain Patch
- Placebo Patch (Placebo Comparator): One Placebo Patch applied once daily for 3 days
  Interventions: Drug: Placebo Patch
- No Treatment (Other): No Treatment for 3 days
  Interventions: Drug: No Treatment

INTERVENTIONS:
Drug: Loxoprofen Pain Patch — One Loxoprofen Pain Patch (active NSAID) applied once daily for 3 days
  Arms: Loxoprofen Pain Patch
Drug: Placebo Patch — One Placebo Patch applied daily for 3 days
  Arms: Placebo Patch
Drug: No Treatment — No Treatment for 3 days
  Arms: No Treatment

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy and safety of a new pain patch compared to placebo and no treatment in subjects experiencing Delayed Onset Muscle Soreness (DOMS).

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 40 years of age
* are in good general health, with a BMI less than or equal to 32, and able to perform the exercise regimen
* develops muscle pain/soreness within 24-48 hours of the end of the exercise regimen and have a baseline muscle pain/soreness with movement of greater than or equal to 5 on the Numerical Rating Scale (NRS) (numerical rating scale) and at least "moderate" on the categorical scale

Exclusion Criteria:

* has engaged in upper extremity exercise for a minimum of 6 months prior to study participation
* has been working heavy manual or physical labor jobs within 3 months prior to study participation.
* has a known history of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, or any nonsteroidal anti-inflammatory drugs
* has skin lesions such as psoriasis at the application site
* has abnormal skin condition such as eczema, contact dermatitis, pigment anomaly, etc.
* has an allergy-related skin condition

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sum of pain intensity differences over 24 hours from baseline (SPID 24) with movement | 0-24 hours

SECONDARY OUTCOMES:
Sum of pain intensity differences over 24 hours from baseline (SPID 24) at rest | 0-24 hours
Sum of pain intensity differences over 48 hours from baseline (SPID 48) with movement | 0-48 hours
Sum of pain intensity differences over 48 hours from baseline (SPID 48) at rest | 0-48 hours
Time to onset of first perceptible pain relief | First 4 hours after Dose 1
Time to onset of meaningful pain relief | First 4 hours after Dose 1
Subjects global impression of medication | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Derek Muse, MD, Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States